CLINICAL TRIAL: NCT01724398
Title: Safety and Efficacy of Human Umbilical Cord Mesenchymal Stem Cells Transplantation Combined With Plasma Exchange for Patients With Acute-on-Chronic Liver Failure Caused by Hepatitis B Virus (HBV)
Brief Title: Umbilical Cord Mesenchymal Stem Cells Transplantation Combined With Plasma Exchange for Patients With Liver Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-PE
Record Dates: First submitted 2012-11-04; First posted 2012-11-09 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Liver Failure
Keywords: mesenchymal stem cells; plasma exchange; liver failure; hepatitis B virus
MeSH Terms: conditions — Liver Failure; Hepatitis B | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Conventional treatment (Experimental): Participants will receive conventional treatment and then be followed until the week 48 study visit.
  Interventions: Other: Conventional treatment
- Conventional plus UC-MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of UC-MSC and then be followed until the week 48 study visit.
  Interventions: Other: Conventional plus UC-MSC treatment
- Conventional plus PE treatment (Experimental): Participants will receive conventional treatment plus plasma exchange and then be followed until the week 48 study visit.
  Interventions: Other: Conventional plus PE treatment
- Conventional plus UC-MSC and PE therapy (Experimental): Participants will receive conventional treatment plus umbilical cord mesenchymal stem cells transplantation combined with plasma exchange. Participants will then be followed until the week 48 study visit.
  Interventions: Other: Conventional plus UC-MSC and PE therapy

INTERVENTIONS:
Other: Conventional plus UC-MSC treatment — Received conventional treatment and umbilical cord mesenchymal stem cells transplantation by peripheral vein slowly for 30minutes. (1×105/Kg, once a week, 4 times).
  Arms: Conventional plus UC-MSC treatment
Other: Conventional plus PE treatment — Received conventional treatment plus 2000 milliliter plasma exchange (every 3 days, 3 times).
  Arms: Conventional plus PE treatment
Other: Conventional plus UC-MSC and PE therapy — Received conventional treatment plus 2000 milliliter plasma exchange (every 3 days, 3 times). Meantime taken i.v umbilical cord mesenchymal stem cells transplantation slowly for 30minutes (1×105/Kg, once a week, 4 times), the first two times is taken after plasma exchange.
  Arms: Conventional plus UC-MSC and PE therapy
Other: Conventional treatment — Received conventional treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Arms: Conventional treatment

SUMMARY:
Liver failure (LF) is a dramatic clinical syndrome with massive necrosis of liver cells. Although liver transplantation provides an option to cure patients suffering with LF, lack of donors, postoperative complications, especially rejection, and high cost limit its application. Previous study showed that bone marrow derived mesenchymal stem cells (BM-MSCs) the novel and promising therapeutic strategy, BM-MSCs can replace hepatocytes in injured liver, and effectively rescue experimental liver failure and contribute to liver regeneration. Plasma exchange (PE) can improve internal environment by removing endotoxin, it helps the liver regeneration and functional recovery and make UC-MSC differentiation into hepatocyte like cells, and exert immunomodulatory function. In this study, safety and efficacy of human umbilical cord mesenchymal stem cells (UC-MSCs) transplantation combined with plasma exchange (PE) for patients with liver failure caused by hepatitis B Virus will be evaluated.

DETAILED DESCRIPTION:
To investigate safety and efficacy of human umbilical cord mesenchymal stem cells (UC-MSCs) transplantation combined with plasma exchange (PE) for patients with liver failure caused by hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Acute-on-Chronic liver failure caused by hepatitis B virus
* Model for End-Stage Liver Disease (MELD) <30

Exclusion Criteria:

* Liver failure caused by other reasons, such as autoimmune diseases, alcohol, drug and so on
* History of severe hepatic encephalopathy or variceal bleeding during the last two months before enrollment
* Severe problems in other vital organs(e.g. the heart, renal or lungs)
* Severe bacteria infection
* Tumor on ultrasonography, CT or MRI examination
* Pregnant or lactating women

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Survival rate and time | 48 weeks

SECONDARY OUTCOMES:
Improve biochemical indexes [alanine aminotransferase (ALT), albumin (ALB), total bilirubin (TBIL), prothrombin time (PT), INR and so on] | 24 weeks after treatment
The clinical symptom improvement [including appetite, debilitation, abdominal distension, edema of lower limbs, et al] | 24 weeks after treatment
Liver function evaluation using Child-Pugh score and MELD score | 24 weeks after treatment
Immune function improvement [including Th1/Th2] | 24 weeks after treatment
The occurrence of complications [including body temperature, tetter and allergy] | Between 0 to 8 hours after UC-MSCs transfusion
Incidence of hepatocellular carcinoma | 48 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Liang Gao, Doctor, Principal Investigator — The Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xu WX, He HL, Pan SW, Chen YL, Zhang ML, Zhu S, Gao ZL, Peng L, Li JG. Combination Treatments of Plasma Exchange and Umbilical Cord-Derived Mesenchymal Stem Cell Transplantation for Patients with Hepatitis B Virus-Related Acute-on-Chronic Liver Failure: A Clinical Trial in China. Stem Cells Int. 2019 Feb 4;2019:4130757. doi: 10.1155/2019/4130757. eCollection 2019. PMID 30863450